CLINICAL TRIAL: NCT00560885
Title: AtriCure Synergy Bipolar RF Energy Lesions for Permanent Atrial Fibrillation Treatment During Concomitant On-Pump Endo/Epicardial Cardiac Surgery
Brief Title: AtriCure Bipolar Radiofrequency Ablation of Permanent Atrial Fibrillation
Acronym: ABLATE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AtriCure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP2007-1
Record Dates: First submitted 2007-11-19; First posted 2007-11-20 (Estimated); Results first posted 2013-03-14 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; af; ablation; arrhythmia; racing heart; afib; surgical ablation
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Tachycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AtriCure Bipolar System (Experimental): The AtriCure Synergy Bipolar Ablation system is used to create lesions outlined in the Maze IV procedure during a concomitant open cardiac surgical procedure.
  Interventions: Device: AtriCure Bipolar System

INTERVENTIONS:
Device: AtriCure Bipolar System — Surgical bipolar radiofrequency ablation using the AtriCure Bipolar System

SUMMARY:
ABLATE is a prospective, non-randomized multi-center clinical trial to demonstrate the safety and effectiveness of the AtriCure Bipolar System for treating permanent atrial fibrillation during concomitant on-pump cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is greater than or equal to 18 years of age
2. Subject has history of permanent atrial fibrillation as defined by the ACC/AHA/ESC Guidelines
3. Subject is scheduled to undergo elective on-pump cardiac surgical procedure(s) for one or more of the following:

   * Mitral valve repair or replacement
   * Aortic valve repair or replacement
   * Tricuspid valve repair or replacement
   * Coronary Artery Bypass procedures
   * Atrial Septal Defect Repair
   * Patent Foramen Ovale closure
4. Subject's Left Ventricular Ejection Fraction ≥ 30%
5. Subject is able and willing to provide written informed consent and comply with study requirements
6. Subject has life expectancy of at least 1 year

Exclusion Criteria:

1. Stand alone AF without indication(s) for concomitant CABG, valve surgery, ASD repair, or PFO closure
2. Previous cardiac ablation including catheter ablation, AV-nodal ablation, or surgical Maze procedure
3. Wolff-Parkinson-White syndrome
4. Prior cardiac surgery (Redo)
5. Class IV NYHA heart failure symptoms
6. Prior history of cerebrovascular accidents within 6 months or at any time if there is residual neurological deficit
7. Documented MI within 6 weeks prior to study enrollment
8. Need for emergent cardiac surgery (i.e. cardiogenic shock)
9. Known carotid artery stenosis greater than 80%
10. LA size greater than or equal to 8cm
11. Current diagnosis of active systemic infection
12. Severe peripheral arterial occlusive disease defined as claudication with minimal exertion
13. Pregnancy or desire to get pregnant within 12-months of the study enrollment
14. Preoperative need for an intra-aortic balloon pump or intravenous inotropes
15. Renal failure requiring dialysis or hepatic failure
16. Requires anti-arrhythmic drug therapy for the treatment of a ventricular arrhythmia
17. Therapy resulting in compromised tissue integrity including: thoracic radiation, chemotherapy, long term treatment with oral or injected steroids, or known connective tissue disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-11; Primary Completion 2009-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Mercy Heart Institute, Sacramento, California
  - Sutter Health, Sacramento, California
  - Heart Center of Indiana, Indianapolis, Indiana
  - Spectrum Health, Grand Rapids, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Baylor Heart Hospital, Dallas, Texas
  - Inova Fairfax, Falls Church, Virginia
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Treatment subjects were recruited from the routine clinical referral base of one or more surgeons at each investigational site.
Pre-assignment Details: Subjects were screened for enrollment and consented prior to being brought to the OR with the potential that they may not be eligible based on some criteria evaluated in OR (i.e. left atrial size assessed by TEE). 1 subject was found to have LA size that excluded them from the trial.
Groups:
- AtriCure Bipolar System: The AtriCure Synergy Bipolar Ablation system is used to create lesions outlined in the Maze IV procedure during a concomitant open cardiac surgical procedure.
  AtriCure Bipolar System : Surgical bipolar radiofrequency ablation using the AtriCure Bipolar System
Period: Overall Study
Arm/Group | AtriCure Bipolar System
Started | 55
30 Day Follow-up | 53 (53 pts available for 30 day follow-up, 52 pts assessed)
3 Month Follow-up | 51 (51 pts available for 3 month follow-up, 48 pts assessed.)
6 Month Follow-up | 50 (50 pts available for 6 month follow-up, 50 pts assessed)
12 Month Follow-up | 48 (48 pts available for 12 month follow-up, 46 pts assessed)
2 Year Follow-up | 47
Completed | 47
Not Completed | 8
Not completed — Death | 7
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | AtriCure Bipolar System
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 43
Age Continuous [Mean (Standard Deviation); unit: years] | 70.5 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 32
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Free From AF and Off Class I and III Anti-arrhythmic Drugs as Determined by Holter Monitoring at 6 Months.
Time Frame: 6 Months Post Procedure
Population: The analysis population included subjects that were evaluable for the Primary Efficacy Endpoint. The completer population excluded 5 subjects. These were 2 post op deaths, 2 deaths beyond 3 months but less than 6 months and 1 subject that withdrew at the 30 day visit.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | AtriCure Bipolar System
Number analyzed (Participants) | 50
percentage of subjects | 74 [60 to 100]

2. Primary Outcome: Composite Acute Major Adverse Event Rate, Within 30 Days Post-procedure or Hospital Discharge
Description: Major Adverse Events consist of Death within 30 days or beyond 30 days if considered device related, Excessive Bleeding, Stroke, TIA or MI. A clinic visist was performed at 30 days to fully assess the patient for adverse events.
Time Frame: 30 days Post Procedure
Population: Safety was evaluated in all subjects enrolled and treated with the device.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | AtriCure Bipolar System
Number analyzed (Participants) | 55
percentage of subjects | 9.1 [0 to 17.9]

3. Secondary Outcome: Percent of Patients Free From AF, Independent of Antiarrhythmic Drug Status as Determined by Holter Monitoring at 6 Months.
Time Frame: 6 Months Post Procedure
Population: The analysis population included subjects that were evaluable for the Secondary Efficacy Endpoint. The completer population excluded 5 subjects. These were 2 post op deaths, 2 deaths beyond 3 months but less than 6 months and 1 subject that withdrew at the 30 day visit.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | AtriCure Bipolar System
Number analyzed (Participants) | 50
percentage of subjects | 84 [66.7 to 94.6]

4. Secondary Outcome: Composite 6-month Post-procedure Major Adverse Event Rate.
Time Frame: 6 Months Post Procedure
Population: Safety was evaluated in all subjects enrolled and treated with the device.
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | AtriCure Bipolar System
Number analyzed (Participants) | 55
percentage of subjects | 10.9 [2.9 to 26.1]

ADVERSE EVENTS:
Time Frame: Primary safety endpoint is rate of Major Adverse Events occuring at 30 days post procedure. Secondary safety endpoint is the composite 6 month post procedure Major Adverse Event rate. Adverse events were collected through 12 month follow up.
Description: Major Adverse Events wre Death, Stroke, Transient Ischemic Attacks, Myocardial infarction and Excessive Bleeding
Arm/Group | AtriCure Bipolar System
Serious Adverse Events (participants affected / at risk) | 45/55
Other Adverse Events (participants affected / at risk) | 51/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AtriCure Bipolar System (N=55)
Anaemia (Blood and lymphatic system disorders) | 4 (4)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Atrial rupture (Cardiac disorders) | 1 (1)
Atrioventricular block (Cardiac disorders) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 8 (8)
Cardiac failure congestive (Cardiac disorders) | 11 (11)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 2 (2)
Mitral valve incompetence (Cardiac disorders) | 2 (2)
Nodal arrhythmia (Cardiac disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 2 (2)
Sick sinus syndrome (Cardiac disorders) | 1 (1)
Sinus arrest (Cardiac disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Sudden death (General disorders) | 1 (1)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (2)
Bacteraemia (Infections and infestations) | 1 (1)
Breast abscess (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 4 (4)
Sepsis (Infections and infestations) | 2 (2)
Wound infection (Infections and infestations) | 1 (1)
Atrial rupture (Injury, poisoning and procedural complications) | 1 (1)
Cardiac procedure complication (Injury, poisoning and procedural complications) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Vena cava injury (Injury, poisoning and procedural complications) | 1 (1)
Venous injury (Injury, poisoning and procedural complications) | 1 (1)
Hyponatraemia (Injury, poisoning and procedural complications) | 1 (1)
Critical illness polyneuropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 7 (7)
Renal mass (Renal and urinary disorders) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 10 (11)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 12 (13)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AtriCure Bipolar System (N=55)
Bradycardia (Cardiac disorders) | 14 (14)
Cardiac Failure Congestive (Cardiac disorders) | 11 (12)
Nodal Arrhythmia (Cardiac disorders) | 3 (3)
Sinus bradycardia (Cardiac disorders) | 5 (5)
Candidiasis (Infections and infestations) | 4 (4)
Pneumonia (Infections and infestations) | 6 (6)
Urinary Tract Infection (Infections and infestations) | 6 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 9 (10)
Renal Failure (Renal and urinary disorders) | 8 (8)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 17 (21)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Haemorrhage (Vascular disorders) | 12 (13)
Hypotension (Vascular disorders) | 3 (3)
Coagulopathy (Blood and lymphatic system disorders) | 5 (5)
Anaemia (Blood and lymphatic system disorders) | 18 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor can review communications prior to public release and can embargo communication regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the tim submitted to the sponsor for review. The sponsor can redact or modify the proposed publication to remove any language the sponsor believes would be detrimental to intellectual property or inaccurately reflect the results of the study.